CLINICAL TRIAL: NCT00693238
Title: A Phase II Study of Hypofractionated Image Guided Proton Radiation Therapy for Low and Intermediate Risk Adenocarcinoma of the Prostate
Brief Title: Proton Therapy for Low and Intermediate Risk Prostate Cancer
Acronym: PR04
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UFPTI 0702-PR04; IRB201701653 (Other: UF IRB); UFJ 2008-022 (Other: UF IRB Old)
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Results first posted 2013-07-24 (Estimated); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Proton Radiation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Risk Proton Radiation (Experimental): 70 Gy/CGE in 28 fractions of 2.5 Gy/CGE/fx
  Interventions: Radiation: Low Risk Proton Radiation
- Intermediate Risk Proton Radiation (Experimental): 72.5 GY/CGE in 29 fractions of 2.5 Gy/CGE/fx
  Interventions: Radiation: Intermediate Risk Proton Radiation

INTERVENTIONS:
Radiation: Low Risk Proton Radiation
  Arms: Low Risk Proton Radiation
Radiation: Intermediate Risk Proton Radiation
  Arms: Intermediate Risk Proton Radiation

SUMMARY:
The purpose of this trial is to give a shorter course (5 ½ weeks) of radiation that has as little side effects on normal bladder and rectal tissues as the usual longer course (8 weeks) of radiation, without decreasing the chance of killing prostate cancer cells.

DETAILED DESCRIPTION:
Low Risk - Total of 70 Gy/CGE over 28 treatments

Intermediate Risk - Total of 72.5 Gy/CGE over 29 treatments

ELIGIBILITY:
Inclusion Criteria

* Prostate cancer.
* Gleason score 2-7.
* PSA ≤ 20 ng/ml.

Exclusion Criteria:

* Previous prostate cancer surgery or pelvic radiation.
* Prior or current chemotherapy for prostate cancer.
* Active inflammatory bowel disease (Crohn's disease, diverticulitis or ulcerative colitis) affecting the rectum.
* History of proximal urethral stricture requiring dilatation.
* History of hip replacement.
* Diabetes requiring medication.
* Prior intrapelvic surgery.
* Current and continuing anticoagulation with Warfarin sodium (Coumadin), Clopidogrel bisulfate (Plavix), enoxaparin sodium (Lovenox), or aspirin/er dipyridamole (Aggrenox).
* On Flomax (Tamsulosin), Hytrin (Terazosin) or Cardura (Doxazosin), Uroxatral (alfuzosin HCl).
* Taking Saw Palmetto or methotrexate and unable or unwilling to discontinue its use during radiation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2008-04; Primary Completion 2012-06 (Actual); Study Completion 2022-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randal H Henderson, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

REFERENCES:
- [Background] American Cancer Society. 2007. Ref Type: Electronic Citation
- [Background] Soloway MS, Pareek K, Sharifi R, Wajsman Z, McLeod D, Wood DP Jr, Puras-Baez A; Lupron Depot Neoadjuvant Prostate Cancer Study Group. Neoadjuvant androgen ablation before radical prostatectomy in cT2bNxMo prostate cancer: 5-year results. J Urol. 2002 Jan;167(1):112-6. PMID 11743286
- [Background] Hull GW, Rabbani F, Abbas F, Wheeler TM, Kattan MW, Scardino PT. Cancer control with radical prostatectomy alone in 1,000 consecutive patients. J Urol. 2002 Feb;167(2 Pt 1):528-34. doi: 10.1016/S0022-5347(01)69079-7. PMID 11792912
- [Background] Kestin LL, Martinez AA, Stromberg JS, Edmundson GK, Gustafson GS, Brabbins DS, Chen PY, Vicini FA. Matched-pair analysis of conformal high-dose-rate brachytherapy boost versus external-beam radiation therapy alone for locally advanced prostate cancer. J Clin Oncol. 2000 Aug;18(15):2869-80. doi: 10.1200/JCO.2000.18.15.2869. PMID 10920135
- [Background] Merrick GS, Butler WM, Wallner KE, Galbreath RW, Allen ZA, Adamovich E. The impact of primary Gleason grade on biochemical outcome following brachytherapy for hormone-naive Gleason score 7 prostate cancer. Cancer J. 2005 May-Jun;11(3):234-40. doi: 10.1097/00130404-200505000-00010. PMID 16053667
- [Background] Demanes DJ, Rodriguez RR, Schour L, Brandt D, Altieri G. High-dose-rate intensity-modulated brachytherapy with external beam radiotherapy for prostate cancer: California endocurietherapy's 10-year results. Int J Radiat Oncol Biol Phys. 2005 Apr 1;61(5):1306-16. doi: 10.1016/j.ijrobp.2004.08.014. PMID 15817332
- [Background] D'Amico AV, Whittington R, Malkowicz SB, Schultz D, Blank K, Broderick GA, Tomaszewski JE, Renshaw AA, Kaplan I, Beard CJ, Wein A. Biochemical outcome after radical prostatectomy, external beam radiation therapy, or interstitial radiation therapy for clinically localized prostate cancer. JAMA. 1998 Sep 16;280(11):969-74. doi: 10.1001/jama.280.11.969. PMID 9749478
- [Background] Common Terminology Criteria for Adverse Events v3.0 (CTCAE). National Cancer Institute. 12-12-0003. 9-9-0005. Ref Type: Electronic Citation
- [Background] Chism DB, Hanlon AL, Horwitz EM, Feigenberg SJ, Pollack A. A comparison of the single and double factor high-risk models for risk assignment of prostate cancer treated with 3D conformal radiotherapy. Int J Radiat Oncol Biol Phys. 2004 Jun 1;59(2):380-5. doi: 10.1016/j.ijrobp.2003.10.059. PMID 15145151
- [Background] Martinez AA, Demanes DJ, Galalae R, Vargas C, Bertermann H, Rodriguez R, Gustafson G, Altieri G, Gonzalez J. Lack of benefit from a short course of androgen deprivation for unfavorable prostate cancer patients treated with an accelerated hypofractionated regime. Int J Radiat Oncol Biol Phys. 2005 Aug 1;62(5):1322-31. doi: 10.1016/j.ijrobp.2004.12.053. PMID 16029788
- [Background] Roach M, Lu J, Pilepich MV, Asbell SO, Mohiuddin M, Terry R, Grignon D. Four prognostic groups predict long-term survival from prostate cancer following radiotherapy alone on Radiation Therapy Oncology Group clinical trials. Int J Radiat Oncol Biol Phys. 2000 Jun 1;47(3):609-15. doi: 10.1016/s0360-3016(00)00578-2. PMID 10837943
- [Background] Ghilezan MJ, Jaffray DA, Siewerdsen JH, Van Herk M, Shetty A, Sharpe MB, Zafar Jafri S, Vicini FA, Matter RC, Brabbins DS, Martinez AA. Prostate gland motion assessed with cine-magnetic resonance imaging (cine-MRI). Int J Radiat Oncol Biol Phys. 2005 Jun 1;62(2):406-17. doi: 10.1016/j.ijrobp.2003.10.017. PMID 15890582
- [Background] Padhani AR, Khoo VS, Suckling J, Husband JE, Leach MO, Dearnaley DP. Evaluating the effect of rectal distension and rectal movement on prostate gland position using cine MRI. Int J Radiat Oncol Biol Phys. 1999 Jun 1;44(3):525-33. doi: 10.1016/s0360-3016(99)00040-1. PMID 10348281
- [Background] Litzenberg D, Dawson LA, Sandler H, Sanda MG, McShan DL, Ten Haken RK, Lam KL, Brock KK, Balter JM. Daily prostate targeting using implanted radiopaque markers. Int J Radiat Oncol Biol Phys. 2002 Mar 1;52(3):699-703. doi: 10.1016/s0360-3016(01)02654-2. PMID 11849792
- [Background] Litzenberg DW, Balter JM, Hadley SW, Sandler HM, Willoughby TR, Kupelian PA, Levine L. Influence of intrafraction motion on margins for prostate radiotherapy. Int J Radiat Oncol Biol Phys. 2006 Jun 1;65(2):548-53. doi: 10.1016/j.ijrobp.2005.12.033. Epub 2006 Mar 20. PMID 16545919
- [Background] Vargas C, Yan D, Kestin LL, Krauss D, Lockman DM, Brabbins DS, Martinez AA. Phase II dose escalation study of image-guided adaptive radiotherapy for prostate cancer: use of dose-volume constraints to achieve rectal isotoxicity. Int J Radiat Oncol Biol Phys. 2005 Sep 1;63(1):141-9. doi: 10.1016/j.ijrobp.2004.12.017. PMID 16111582
- [Background] Vargas C, Martinez A, Kestin LL, Yan D, Grills I, Brabbins DS, Lockman DM, Liang J, Gustafson GS, Chen PY, Vicini FA, Wong JW. Dose-volume analysis of predictors for chronic rectal toxicity after treatment of prostate cancer with adaptive image-guided radiotherapy. Int J Radiat Oncol Biol Phys. 2005 Aug 1;62(5):1297-308. doi: 10.1016/j.ijrobp.2004.12.052. PMID 16029785
- [Background] Dearnaley DP, Hall E, Lawrence D, Huddart RA, Eeles R, Nutting CM, Gadd J, Warrington A, Bidmead M, Horwich A. Phase III pilot study of dose escalation using conformal radiotherapy in prostate cancer: PSA control and side effects. Br J Cancer. 2005 Feb 14;92(3):488-98. doi: 10.1038/sj.bjc.6602301. PMID 15685244
- [Background] Pollack A, Zagars GK, Starkschall G, Antolak JA, Lee JJ, Huang E, von Eschenbach AC, Kuban DA, Rosen I. Prostate cancer radiation dose response: results of the M. D. Anderson phase III randomized trial. Int J Radiat Oncol Biol Phys. 2002 Aug 1;53(5):1097-105. doi: 10.1016/s0360-3016(02)02829-8. PMID 12128107
- [Background] Sathya JR, Davis IR, Julian JA, Guo Q, Daya D, Dayes IS, Lukka HR, Levine M. Randomized trial comparing iridium implant plus external-beam radiation therapy with external-beam radiation therapy alone in node-negative locally advanced cancer of the prostate. J Clin Oncol. 2005 Feb 20;23(6):1192-9. doi: 10.1200/JCO.2005.06.154. PMID 15718316
- [Background] Shipley WU, Verhey LJ, Munzenrider JE, Suit HD, Urie MM, McManus PL, Young RH, Shipley JW, Zietman AL, Biggs PJ, et al. Advanced prostate cancer: the results of a randomized comparative trial of high dose irradiation boosting with conformal protons compared with conventional dose irradiation using photons alone. Int J Radiat Oncol Biol Phys. 1995 Apr 30;32(1):3-12. doi: 10.1016/0360-3016(95)00063-5. PMID 7721636
- [Background] Vargas, C, Martinez, A, and Boike, T. Long term survival benefit of a prospective dose escalation trial using high dose rate (HDR) brachytherapy boost. Int.J.Radiat.Oncol.Biol.Phys.2005. Ref Type: Abstract
- [Background] Vargas C, Martinez A, Galalae R, Demanes J, Harsolia A, Schour L, Nuernberg N, Gonzalez J. High-dose radiation employing external beam radiotherapy and high-dose rate brachytherapy with and without neoadjuvant androgen deprivation for prostate cancer patients with intermediate- and high-risk features. Prostate Cancer Prostatic Dis. 2006;9(3):245-53. doi: 10.1038/sj.pcan.4500882. Epub 2006 Jun 20. PMID 16786040
- [Background] Zietman AL, DeSilvio ML, Slater JD, Rossi CJ Jr, Miller DW, Adams JA, Shipley WU. Comparison of conventional-dose vs high-dose conformal radiation therapy in clinically localized adenocarcinoma of the prostate: a randomized controlled trial. JAMA. 2005 Sep 14;294(10):1233-9. doi: 10.1001/jama.294.10.1233. PMID 16160131
- [Background] Kupelian PA, Reddy CA, Klein EA, Willoughby TR. Short-course intensity-modulated radiotherapy (70 GY at 2.5 GY per fraction) for localized prostate cancer: preliminary results on late toxicity and quality of life. Int J Radiat Oncol Biol Phys. 2001 Nov 15;51(4):988-93. doi: 10.1016/s0360-3016(01)01730-8. PMID 11704322
- [Background] Kupelian PA, Reddy CA, Carlson TP, Altsman KA, Willoughby TR. Preliminary observations on biochemical relapse-free survival rates after short-course intensity-modulated radiotherapy (70 Gy at 2.5 Gy/fraction) for localized prostate cancer. Int J Radiat Oncol Biol Phys. 2002 Jul 15;53(4):904-12. doi: 10.1016/s0360-3016(02)02836-5. PMID 12095556
- [Background] Kupelian PA, Thakkar VV, Khuntia D, Reddy CA, Klein EA, Mahadevan A. Hypofractionated intensity-modulated radiotherapy (70 gy at 2.5 Gy per fraction) for localized prostate cancer: long-term outcomes. Int J Radiat Oncol Biol Phys. 2005 Dec 1;63(5):1463-8. doi: 10.1016/j.ijrobp.2005.05.054. Epub 2005 Sep 19. PMID 16169683
- [Background] Slater JD, Rossi CJ Jr, Yonemoto LT, Bush DA, Jabola BR, Levy RP, Grove RI, Preston W, Slater JM. Proton therapy for prostate cancer: the initial Loma Linda University experience. Int J Radiat Oncol Biol Phys. 2004 Jun 1;59(2):348-52. doi: 10.1016/j.ijrobp.2003.10.011. PMID 15145147
- [Derived] Henderson RH, Bryant C, Hoppe BS, Nichols RC, Mendenhall WM, Flampouri S, Su Z, Li Z, Morris CG, Mendenhall NP. Five-year outcomes from a prospective trial of image-guided accelerated hypofractionated proton therapy for prostate cancer. Acta Oncol. 2017 Jul;56(7):963-970. doi: 10.1080/0284186X.2017.1287946. Epub 2017 Feb 22. PMID 28514929
- See also: Contact the University of Florida Proton Therapy Institute — https://www.floridaproton.org/about-us/contact-us

RESULTS

PARTICIPANT FLOW:
Recruitment Details: University of Florida Proton Therapy Institute, between 04/2008 and 04/2010
Period: Overall Study
Arm/Group | Low Risk Proton Radiation | Intermediate Risk Proton Radiation
Started | 122 | 106
Completed | 122 | 106
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Risk Proton Radiation | Intermediate Risk Proton Radiation | Total
Number analyzed (Participants) | 122 | 106 | 228
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 60 | 44 | 104
  >=65 years | 62 | 62 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (7.5) | 64.1 (6.9) | 64.7 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 122 | 106 | 228
Region of Enrollment [Number; unit: participants]
  United States | 122 | 106 | 228

OUTCOME MEASURES:

1. Primary Outcome: Acute Grade 3 (NCI CTC v4.0) or Higher Treatment-related Toxicity Rate.
Time Frame: 6 months after the end of radiation therapy
Measure: Number; unit: Participants
Arm/Group | Low Risk Proton Radiation | Intermediate Risk Proton Radiation
Number analyzed (Participants) | 122 | 106
Participants | 0 | 0

2. Secondary Outcome: Disease Control
Time Frame: 20 years after end of radiation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: These serious events cover the range from during treatment to the maximum available follow-up for any given patient (current maximum of 4.5 years).
Arm/Group | Low Risk Proton Radiation | Intermediate Risk Proton Radiation
Serious Adverse Events (participants affected / at risk) | 2/122 | 2/106
Other Adverse Events (participants affected / at risk) | 26/122 | 21/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Risk Proton Radiation (N=122) | Intermediate Risk Proton Radiation (N=106)
Rectal hemmorhage (grade 3) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctitis (grade 3) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary retention (grade 3) (Renal and urinary disorders) | 1 (1) | 0 (0)
Hematuria (grade 3) (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Risk Proton Radiation (N=122) | Intermediate Risk Proton Radiation (N=106)
Rectal hemmorhage (Gastrointestinal disorders) | 12 (12) | 14 (14)
Urinary Frequency/urgency (Renal and urinary disorders) | 22 (22) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes